CLINICAL TRIAL: NCT06809244
Title: Strength Training for Persons with Eating Disorders: a Pilot Study
Brief Title: Strength Training and Eating Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: Modum Bad (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Solfrid Bratland Sanda, Professor, University of South-Eastern Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STRENGTHANDED_PILOT
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders
Keywords: exercise; eating disorders; affective responses
MeSH Terms: conditions — Feeding and Eating Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Strength training (Experimental): Perform one maximal strength training session (5RM x 3 sets) and one hypertrophy strength training session (10RM x 3 sets). Both sessions include 5 exercises (squat or leg press, bench press or chest press, deadlift, lounges and pull-down)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Strength training as described under "arm"

SUMMARY:
The aim of this pilot study is to test feasibility of assessment methods and immediate responses to two different strength training sessions, maximal strength training and hypertrophy strength training, among persons undergoing treatment for eating disorders. The study will combine quantitative methods to assess immediate physiological and affective responses to two adapted and supervised strength training sessions. Following the sessions, qualitative in-dept interviews will address the participants' experiences with the strength training sessions. A total of 30 participants from different treatment settings for eating disorders will be recruited to participation. Assessments include symptoms of eating disorders, muscle strength, physical activity behaviour and motivation, blood pressure, heart rate variability, body temperature, lactate, percievied exertion and affective responses. The findings of the study will be utilized in a randomized clinical trial with strength training as part of treatment for eating disorders.

DETAILED DESCRIPTION:
Eating disorders are widespread mental disorders with a social cost of approximately NOK 26 billion per year (Streatfeild et al., 2021), and which are characterised by a long duration, high level of suffering and a very negative impact on quality of life (Hay et al., 2023). Despite good research-based documentation of effective treatments for eating disorders, approximately one-third of people undergoing treatment for eating disorders experience no improvement (Vrabel et al., 2008).

Maladaptive physical activity and exercise, i.e. exercise that results in a negative impact on health and quality of life, is a common symptom in many people with eating disorders, and it has been particularly documented for people with Anorexia Nervosa and Bulimia Nervosa (Gorrell et al., 2021; Quesnel et al., 2023). This symptom predicts longer treatment time, poorer treatment outcomes and an increased risk of relapse (Strober et al., 1997). Various attempts have been made to manage this type of exercise, and for a long time the prevailing paradigm was that this was best managed with bed rest (Ibrahim et al., 2019). This is similar to the paradigms from the early and mid-20th century for convalescence after, for example, myocardial infarction (André, 2020), but where physical activity was experimented with in the 1960s and where the treatment regime has evolved to now recommend high-intensity endurance training and limiting bed rest and sedentary behaviour (Bahr, 2009).

Several case studies have shown that maximal strength training as part of treatment is feasible for people with anorexia nervosa (Bratland-Sanda et al., 2018; Healy et al., 2024), while other studies have found the effect of strength training with more repetitions and lower load on both adolescents and adults with anorexia nervosa (Fernandez-Del-Valle, Larumbe-Zabala, Morande-Lavin, et al., 2015; Fernandez-del-Valle et al., 2014). A clinical study from Norway also showed effects of maximal strength training in the treatment of Bulimia Nervosa and binge eating disorder (Mathisen et al., 2018; Mathisen et al., 2017), and that participants experienced both the content of the training and the meeting with competent, training professionals as useful and important (Bakland et al., 2019).

A recently published scoping review showed that the knowledge gaps for exercise as part of treatment for eating disorders lie particularly in the immediate physiological and affective responses to different forms of exercise and the effects of more systematic use of competent exercise professionals for guidance and follow-up of exercise (Mathisen et al., 2023). There is also a great need for knowledge about how different forms of strength training are experienced by people with eating disorders and different clinical settings, such as inpatient treatment, day programmes and outpatient treatment.

Goals and issues

The aim of the study is twofold. We want to generate knowledge about A) Immediate physiological and affective responses to strength training in people undergoing treatment for various forms of eating disorders B) Feasibility of strength training in different treatment settings for different forms of eating disorders.

The following research questions are formulated:

1. What physiological responses occur during and after one session of maximal strength training and one session of hypertrophic strength training in individuals undergoing treatment for various forms of eating disorders?
2. What affective responses occur during and after one session of maximal strength training and one session of hypertrophic strength training in people undergoing treatment for various forms of eating disorders?
3. What is the feasibility of maximal strength training and hypertrophic strength training sessions as part of treatment for different forms of eating disorders?
4. How is maximal strength training compared to hypertrophic strength training experienced by people undergoing treatment for various forms of eating disorders?
5. What kind of counselling and follow-up do people with different forms of eating disorders need before, during and after maximal strength training and hypertrophic strength training in a treatment context?

Methodology In this study, an experimental design will be used with the collection of both quantitative and qualitative data.

Participants The sample will consist of individuals who fulfil the DSM-5 criteria for the eating disorders Anorexia Nervosa, Bulimia Nervosa, binge eating disorder and unspecified eating disorders (APA, 2013). Individuals will be recruited from the Department of Eating Disorders at Modum Bad, the inpatient department at Lovisenberg Diaconal Hospital, and from outpatient treatment programmes in the public or private sector specifically aimed at eating disorders.

Inclusion criteria:

* Age >18 years
* Under treatment for eating disorders

Exclusion criteria:

* BMI <15 kg/m2
* Established osteoporosis (t-score < -2.5 including low energy fracture)
* Psychosis
* Active suicidality
* Extensive self-harm that interferes with treatment
* Unstable somatic condition

Power calculation This pilot study will be based on both quantitative and qualitative data. As the study has a qualitative approach to investigate experiences with two different types of strength training, and it is not a goal of the study to investigate the effects of the training, we have taken Whitehead et al (2016) as a starting point for calculating the number of participants in the study. This recommends 30 participants in each group for intervention and control groups.In this study, there will only be one intervention group, and with only two sessions in the intervention, the dropout rate will probably be more limited than with a longer intervention period.

We will therefore endeavour to recruit 30 participants. We will endeavour to ensure that the various forms of eating disorders are represented among the participants. Experience indicates that there is a higher proportion of people with unspecified eating disorders, Anorexia Nervosa and Bulimia Nervosa at the two departments that treat eating disorders at Modum Bad and Lovisenberg Diaconal Hospital. We will therefore endeavour to ensure that participants recruited through private clinics also include people with binge eating disorder.

Design and procedure The study will be carried out as an experimental cross-over design in which the participants will be randomised as to which session they start with and which they complete last. All participants will perform one session of maximal strength training, i.e. strength training with heavier and fewer repetitions and with longer breaks between each set, and one hypertrophy strength training, i.e. strength training specifically designed for muscle growth.

The strength training sessions will be carried out at least one week apart to ensure that the sessions do not affect each other.

The following criteria have been established for cancelling participation in the intervention:

* Weight loss greater than 3kg in one week in people with BMI <18.5 kg/m2 and/or
* Physical injury that prevents completion of the strength exercises and/or
* Self-reported emotional discomfort that is directly related to the strength training sessions and is perceived as unmanageable by the participant The weight criterion is assessed through the scheduled weigh-in, physical injury and unmanageable emotional discomfort are assessed through questions and self-report.

Intervention The strength training sessions will be conducted with a warm-up and five full-body exercises using the equipment available at the specific hospital/treatment centre. The warm-up procedure will be standardised. Participants should warm up for a maximum of 15 minutes and the intensity of the warm-up should be low to moderate. It is recommended that participants are allowed to cycle/walk for approximately 10 minutes and then perform a warm-up series of each of the strength exercises.

The exercises to be performed are squat/leg press, bench press/chest press, pull downs, lunges and deadlifts. The exercises will be performed with weights or equipment depending on access. In the maximum strength training session, each exercise will be performed as five repetitions of 5RM x 3 series with at least 2.5 minutes break between each series. In the hypertrophy strength training session, each exercise will be performed as 10 repetitions of 10RM x 3 sets with at least 1 min break between sets.

All the participants will be followed up by an instructor/sports pedagogue during the training sessions throughout the intervention period. This is done both to check attendance and to guide participants on the correct technique and intensity. The instructor must have formal expertise in strength training, and we want to ensure that the instructor has expertise in training guidance for people with eating disorders.

Both compliance (number of sessions completed) and any side effects of the strength training should be recorded.

Measurement of outcome variables We will collect background data on participants' muscle strength and power development, physical activity behaviour, diagnosis, height and weight before the first session.

Muscle strength and power development. 1RM is measured by leg presses and seated chest presses in a machine, power will be measured in the warm-up lifts (maximum mobilisation in the concentric phase). A force platform/muscle lab is used to measure force development (both power and rate of force development).

Physical activity behaviour. Volume (i.e. duration, intensity and frequency) and type of physical activity are self-reported via a training diary; intensity is indicated according to Borg's 6-20 scale (Borg, 1982).Motivation for physical activity is measured via the Behavioural Regulation of Exercise Questionnaire (BREQ-2) (Murcia et al., 2007), while compulsive physical activity is measured via the Compulsive Exercise Test (CET) (Taranis et al., 2011).

Height and weight.We will measure height before the first exercise session, and body weight will be measured before both exercise sessions.

Prior to each of the two sessions, we will collect data on symptoms of eating disorders via the EDE-Q version adapted for frequent measurements (Vrabel et al., 2024). Before, during and after each of the two sessions, we will collect data on physiological and affective responses.

Physiological responses. Blood pressure during and after one strength training session will be measured using a continuous blood pressure monitor (Tango, SunTech, USA). Heart rate, heart rate variability and body temperature will also be measured continuously throughout the sessions using a Polar s610 heart rate monitor (Kempele, Finland) and Oura ring (Oura Health Oy, Oulu, Finland). We will use anonymous user profiles for the Oura rings so that no personally identifiable information is stored by the manufacturer. Data transferred from the manufacturer will be stored on a secure server at Modum Bad. Lactate will be measured during and after each session using a BIOSEN C-line lactate analyser (Biosen, EKF Industrial Electronics, Magdeburg, Germany).

Affective responses. Before, during and after each session, perceived exertion will be self-reported via Borg's scale (Borg, 1982; Kilpatrick et al., 2009), affective responses during the sessions will be measured with the Self-assessment manikin rating scale (SAM) (Bradley & Lang, 1994) and visual analogue scale (VAS) with separate scales for tension, irritation, fatigue, satisfaction and motivation developed after Saanijoki et al. (2015). Affects before and after the sessions will be measured with the Positive and Negative Affect Schedule (PANAS) (Crawford & Henry, 2004; Watson et al., 1988).

Experiences with the training. Qualitative in-depth interviews will be conducted with the participants following the strength training sessions. In this interview, the participants' experiences of the two strength training sessions, the choice of exercises, as well as the guidance and follow-up before, during and after the training session will be thematised. We will also discuss the participants' views on the need for a larger, randomised controlled trial of strength training in the treatment of eating disorders.

Analysis of data We will use statistical analyses with the program SPSS version 29 to describe the data material. This will be done through frequency distribution, mean, standard deviation and confidence intervals. Differences between the two sessions will be analysed using the dependent t-test. The significance level is set at 0.05. In order to analyse the qualitative interviews, a thematic content analysis (Braun & Clarke, 2006) will be conducted on the transcripts of the interviews.

Ethical considerations and considerations The project will fulfil the intentions and conditions of the Health Research Act and the Declaration of Helsinki. The project will be initiated once it has been approved by the Regional Committee for Medical and Health Research Ethics, as well as SIKT and the local data protection officers for research at Modum Bad and Lovisenberg Diakonal Hospital.

'The study can contribute to new knowledge about the response to and experience of two different forms of strength training among people with eating disorders.This is important knowledge when a larger clinical study is to be conducted.All possible adverse events during and after the sessions will be recorded and used in a knowledge base for the development of a clinical study in the area.

The project will fulfil the intentions and conditions of the Health Research Act and the Declaration of Helsinki. The project will be initiated once it has been approved by the Regional Committee for Medical and Health Research Ethics, as well as SIKT and the local data protection officers for research at Modum Bad and Lovisenberg Diakonal Hospital.

The study can contribute to new knowledge about the response to and experience of two different forms of strength training among people with eating disorders. This is important knowledge when conducting a larger clinical study. All possible adverse events during and after the sessions will be recorded and used in a knowledge base for the development of a clinical study in the area.

Data will be collected and stored on a de-identified server at USN.

Assessment of risk of symptom exacerbation and risk of relapse Two sessions should be conducted per participant, with sessions conducted one week apart.Among the acute responses may be that the soreness participants may feel after the sessions will exacerbate concerns about body shape and/or body weight. This can be particularly challenging for people with a high level of body dissatisfaction and who, through their eating disorder, try to switch off and not feel their own body.The questions in the questionnaire and in the interview can also trigger thoughts that may be perceived as demanding.

This will be taken care of by ensuring that all participants are in a defined course of treatment where they have therapists with specialised expertise in eating disorders, and who can thus discuss this with the participants.

Based on previous studies, no adverse events have been reported from longer interventions in this patient group with customised strength training supervised by skilled exercise professionals, i.e. physiotherapists with specific exercise expertise and/or clinical exercise physiologists/sports educators (Bakland et al, 2019; Bratland-Sanda et al, 2018; Fernandez-del-Valle, Larumbe-Zabala, Graell-Berna, et al, 2015; Fernandez-Del-Valle, Larumbe-Zabala, Morande-Lavin, et al, 2015; Fernandez-del-Valle et al, 2014; Healy et al, 2024; Mathisen et al, 2018; Mathisen et al, 2017).

Anecdotally, the collective experience of the clinics included in the project also suggests that the response to such interventions is positive from participants.

While we recognise that there may be a risk that two such sessions may exacerbate the symptoms of the eating disorders regardless of the type of eating disorder diagnosis, it is important to distinguish between increased symptom pressure because a key element of the disorder is addressed, and general relapse of the disease.

For the participants, working on how they relate to exercise in a sustainable way through counselling may create strong reactions, but it is addressed and dealt with in a safe treatment context with experienced and expert therapists.

We will therefore also use our clinical experience of treating various forms of eating disorders, both with and without compulsive exercise as a symptom, to help the participants create an open dialogue about this instead of not addressing it. This is already being done as an ordinary part of treatment at the included clinics, and in this work it is also important to distinguish between what are reactions because the patient is working through something difficult, and what are signs of relapse.

Based on previous studies and clinical experience in the project group, we would assume that the risk for participants is greater in people who have restrictive anorexia with excessive and/or compulsive exercise.

Measures for all participants who experience discomfort and worsening symptoms, regardless of diagnosis, is that this is addressed in the therapy room with the participant's therapist.

If the individual therapist needs guidance on how this can be thematised by the project group's experienced and highly competent psychological specialists, they will receive guidance on this.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing treatment for eating disorders

Exclusion Criteria:

* BMI <15 kg/m2
* established osteoporosis
* psychosis
* active suicidality
* comprehensive self injury behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Participant experiences | 1-3 weeks after performing the two strength training sessions
  Assessed through qualitative in-depth interview

SECONDARY OUTCOMES:
Heart Rate | Measurement during the two 60-min sessions in the intervention
  Heart rate during sessions
Affect | Immediately before and after each of the two 60-minutes strength training sessions
  Positive and Negative Affect Scale (two scores, higher score means greater affect for both postive and negative affects)
Lactate | Immediately before and after each of the three sets of the squat or leg press exercise during the two strength training sessions
  Blood lactate obtained from finger
Affect | Immediately before and after each of the two 60-minutes strength training sessions
  Visual Analogue Scale of tension, motivation, boredom, exitement

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Lovisenberg DIaconal Hospital, Oslo
  - Modum Bad, Vikersund

IPD SHARING:
Plan to Share IPD: Undecided
The sensitivity of the data and the lack of such approval from the ethical committee